CLINICAL TRIAL: NCT05784740
Title: Precision Exercise to Improve Patient Outcomes in Sepsis Survivors: PRECISE Study
Brief Title: Precision Exercise to Improve Outcomes in Sepsis
Acronym: PRECISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other); Simon Fraser University (Other); St. Paul's Hospital, Canada (Other); Providence Health & Services (Other)
Responsible Party: Principal Investigator, Graeme Koelwyn, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H22-02879
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Sepsis
Keywords: Sepsis; Exercise Tolerance; Exercise Training
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Intervention (Experimental): Patients will participate in a 12-week (36 sessions) precision exercise training intervention
  Interventions: Other: 12-week precision exercise training
- Attention Control (No Intervention): Patients will not receive exercise training but will be contacted 1x per week via phone to document self-reported physical activity and general wellbeing.

INTERVENTIONS:
Other: 12-week precision exercise training — The 12-week exercise intervention will consist of both aerobic and strength exercise training performed 3x per week using an individualized and nonlinear periodized approach.
  Arms: Exercise Intervention

SUMMARY:
The goal of this interventional clinical research study is to assess the efficacy of a 12-week precision exercise training intervention to improve exercise tolerance in sepsis survivors.

The main question it aims to answer is does a 12-week precision exercise training program improve constant load exercise time in sepsis survivors?

Participants will:

* Answer questionnaires related to patient reported outcomes and give a blood sample
* Perform a constant load exercise test
* Complete 12-weeks (3 x per week, 36 session in total) of precision exercise training consisting of individualized, nonlinear periodized strength and aerobic exercise training.

Researchers will compare the exercise group to an attention control group of sepsis survivors who do not receive exercise training but instead undergo usual care procedures and receive general lifestyle advice 1x per week.

DETAILED DESCRIPTION:
Sepsis is a life threatening condition that results in multi-organ system dysfunction. In those who survive sepsis, many patients present with chronic immune dysregulation (i.e., paradoxical hyperinflammation and immune suppression), leading to high rates of re-hospitalization. In addition, exercise tolerance is significantly reduced both acutely post hospital discharge and long term (~5 years post initial infection). Exercise training is a pleiotropic intervention that has been demonstrated to improve exercise tolerance in a multitude of clinical populations. Aerobic exercise training is also associated with anti-inflammatory and immune-enhancing effects; however, the magnitude of these immunological adaptations is largely dependent on the exercise prescription used. To date, exercise training studies in sepsis have used a more traditional generic linear exercise training approach, which has resulted in minimal or no effect on exercise tolerance. This is in contrast to other clinical populations wherein precision exercise training (e.g., individualized, nonlinear periodized, combined aerobic and strength training) has resulted in greater improvements in exercise tolerance compared to non-specific linear exercise programs, and is considered safe and tolerable. To date, no study has sought to investigate the effects of a precision exercise training intervention on exercise tolerance and immune function in sepsis survivors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* At least 19 years of age
* ≥60 days prior to study enrollment, known or suspected infection that includes at least two of the following clinical criteria that together constitute a new bedside clinical score termed quickSOFA (qSOFA): respiratory rate >22breaths/min, altered mentation, or systolic blood pressure <100mmHg.
* Cardiorespiratory fitness <80% of age and sex-predicted norms
* Can commit to attending 3 exercise sessions a week for 12-weeks

Exclusion Criteria:

* Unable to provide informed consent
* On supplemental oxygen
* Known previous cardiac or cerebral vascular events in the past 90 days
* Diabetes
* Autoimmune diseases or on daily immunomodulatory drugs
* Obstructive sleep apnea
* Uncontrolled hypertension
* Known pregnancy/ intending to get pregnant within 28 days of enrolling in the study or breastfeeding
* Desaturation during exercise SpO2<85%
* Cardiovascular contraindication or musculoskeletal limitations to exercise as assessed during the cardiopulmonary exercise test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in constant load exercise time | 12-weeks
  Individuals will complete a constant-load exercise trial to symptom limitation at ~70% workload maximum (determined by a cardiopulmonary exercise test) on a cycle ergometer pre to post 12-weeks of the intervention period. The primary outcome will be change in time from pre to post test.

SECONDARY OUTCOMES:
Change in health related quality of life (SF-36) | 12-weeks
  The change in health related quality of life measured by the SF-36 component scores pre to post 12-weeks of the intervention period. The SF 36 Medical Outcomes Study Survey (SF-36) is a 36-item survey that measures quality of life over eight domains, including physical functioning, bodily pain, limitations due to physical health problems, limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. Pre-coded numeric values are assigned to each scale, with items scored from 0-100. High scores represent a more favourable health state. Items in each domain are also averaged to create eight separate domain scores.

OTHER OUTCOMES:
Change in clinical biomarkers of immune function (highly sensitive C-reactive protein) | 12-weeks
  The change in highly sensitive C-reactive protein (mg/L) pre to post 12-weeks of the intervention period.
Change in clinical biomarkers of immune function (absolute lymphocyte count) | 12-weeks
  The change in absolute lymphocyte count (per mL) pre to post 12-weeks of the intervention period.
Change in clinical biomarkers of immune function (monocyte HLA-DR) | 12-weeks
  The change in monocyte human leukocyte antigen-DR (per cell) pre to post 12-weeks of the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Koelwyn, PhD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital - Centre for Heart Lung Innovation, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available as required by a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after publication and for up to 36 months post publication
Access Criteria: The investigator who proposed to use the data and upon reasonable request. Requests should be directed to graeme.koelwyn@hli.ubc.ca. To gain access, data requestors will need to sign a data access agreement.